CLINICAL TRIAL: NCT04626765
Title: An Open, Uncontrolled, Multicenter Clinical Trial to Explore the Safety, Efficacy, and Remission Phase of Chimeric Antigen Receptor T Cell (CAR-T) in the Treatment of Children With Relapsed and Refractory Acute Lymphoblastic Leukemia
Brief Title: CAR-T for Children With Relapsed and Refractory Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T for Childhood B-ALL
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; Influenza Vaccines; Cyclophosphamide; Cholestanetriol 26-Monooxygenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- volunteer (Experimental): The child's parents or legal guardians voluntarily signed the informed consent form, and the child himself/herself met the enter criteria for the diagnosis of patients with acute B-lymphoblastic leukemia (B-ALL) expressing specific target antigens
  Interventions: Drug: CD19 CAR-T; Drug: CD22 CAR-T; Drug: CD 19+22; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: CD19 CAR-T — CD19 CAR-T infusion for pediatric patients with CD19 positive tumor cells
  Other Names: Senl_19
Drug: CD22 CAR-T — CD22 CAR-T infusion for pediatric patients with CD22 positive tumor cells
  Other Names: Senl_22
Drug: CD 19+22 — CD19+22 CAR-T infusion for pediatric patients with CD19 positive and CD22 positive tumor cells
  Other Names: Senl_19+22
Drug: Fludarabine — 25mg/㎡ for D-4、D-3 and D-2
  Other Names: flu
Drug: Cyclophosphamide — 500mg/㎡ for D-3 and D-2
  Other Names: ctx

SUMMARY:
In this study, CAR-T will be administered to children with acute lymphoblastic leukemia to explore the effect of CAR-T intervention time on the duration of complete remission and further verify the long-term safety and efficacy of CAR-T treatment.

DETAILED DESCRIPTION:
After clinician evaluation, if the child meets the study criteria and after adequate communication, the parent or legal guardian voluntarily joins the clinical study, CAR-T technique can be used for related treatment, and the long-term therapeutic effect can be observed. In this trial, 50 children were publicly enrolled and treated with CAR-T. Patients participating in the clinical trial will be tested and assessed in terms of treatment safety, efficacy, and duration of response.

ELIGIBILITY:
Inclusion criteria：

1. The treat history meeting the following criteria:

   Recurrence of lymphoma patients with imaging (CT/MRI/PET-CT) detection and pathological diagnosis, or recurrence including bone marrow morphology relapse and the MRD recurrence of myeloma patients or leukemia patients, after chemotherapy or stem cell transplantation; Can't get complete remission (including MRD positive) after more than twice repeated chemotherapy of incipient lymphoma, myeloma or leukemia patients; One or twice chemotherapy cannot get remission again (including MRD positive), but not suitable for chemotherapy of incipient lymphoma, myeloma or leukemia patients.
2. There is a measurable lesions before treatment at least;
3. ECOG score≤2;
4. To be aged 1 to 18 years;
5. More than a month lifetime from the consent signing date

Exclusion Criteria:

1. Serious cardiac insufficiency, left ventricular ejection fraction<50%;
2. Has a history of severe pulmonary function damaging;
3. Merging other progressing malignant tumor;
4. Merging uncontrolled infection;
5. Merging the metabolic diseases (except diabetes);
6. Merging severe autoimmune diseases or immunodeficiency disease;
7. Patients with active hepatitis B or hepatitis C;
8. Patients with HIV infection;
9. Has a history of serious allergies on Biological products (including antibiotics);
10. Has acute GvHD on allogeneic hematopoietic stem cell transplantation patients after stopping immunosuppressants a month;
11. Any situation that would increase dangerousness of subjects or disturb the outcome of the clinical study according to the researcher's evaluation.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Severe/Adverse Events | 28 days
  Number of Participants with Severe/Adverse Events as a Measure of Safety diagnosis
CAR-T Cell expansion level | 24 months
  Copies numbers of CAR in peripheral blood(PB) and/or bone marrow(BM)

SECONDARY OUTCOMES:
Objective response rate of complete remission and partial remission | 24 months
  Objective response rate of complete remission and partial remission
Overall survival time | 24 months
  Overall survival time

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Luo, PhD&MD, Principal Investigator — The Second Hospital of Hebei Medical University
Locations (1):
- No.2 Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No